CLINICAL TRIAL: NCT07160777
Title: A Single Center Study Evaluating The Clinical Performance and Safety of Hyaluronic Acid-Based Implantable Dermal Fillers Applied to the Face
Brief Title: Performance and Safety of Semical Dermal Fillers in Facial Rejuvenation
Acronym: SEMDERMA
Status: Active, not recruiting | Type: Observational
Sponsor: Semikal Technology (Industry)
Responsible Party: Sponsor
Other Study IDs: SEMDERMA
Record Dates: First submitted 2025-08-15; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Facial Aging; Skin Rejuvenation; Volume Defects in the Mid-face; Lip Augmentation and Correction of Perioral Rhytids; Marionette Lines; Nasolabial Fold Correction; Periorbital Wrinkles; Facial Wrinkles and Rhytides Reduction
Keywords: SEMDERMA; dermal filler; mesolifter; wrinkle correction; lip augmentation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cross-linked Hyaluronic Acid Dermal Filler: Products:
  Semical Dermal Filler- Fine Semical Dermal Filler - Plus Semical Dermal Filler - Ultra
  Cross-linked hyaluronic acid injection for wrinkle correction and/or reshaping of nasolabial folds, marionette lines, crow's feet, perioral lines, periorbital lines, cheek and lip augmentation
  Interventions: Device: cross-linked hyaluronic acid
- Stabilized Non Cross-linked Hyaluronic Acid Mesolifter: Semical Mesolifter injection for rejuvenation and revitalization of facial skin
  Interventions: Device: Mesolifter

INTERVENTIONS:
Device: cross-linked hyaluronic acid — Semical Dermal Filler Fine Semical Dermal Filler Plus Semical Dermal Filler Ultra
  Other Names: Dermal Filler; Hyaluronic acid dermal filler
  Groups: Cross-linked Hyaluronic Acid Dermal Filler
Device: Mesolifter — Stabilized hyaluronic acid with NONASEM Technology. Application with Multi-Aesthetic Point Technique (MAPs)
  Other Names: Skin booster
  Groups: Stabilized Non Cross-linked Hyaluronic Acid Mesolifter

SUMMARY:
The aim of the study is to verify safety and performance of Semical dermal fillers according to real-world data.

DETAILED DESCRIPTION:
This study is a single-center, open label clinical follow-up study. The records of volunteers who were treated with Semical brand dermal fillers on the face at the research center and whose photographs are keps in the researcher's records will be evaluated retrospectively by the principle investigator and an independent evaluator.

Volunteers who were used in accordance with the current intended use declared by the manufacturer of Semical Fine, Plus, Ultra Dermal Fillers and Mesolifter as applied in routine practice by the researcher may be included.

The dermal filler application must have been applied to the necessary and determined facial areas, expectations, product safety requirements, and skin structure, with the technique deemed appropriate by the researcher. In order to obtain optimal aesthetic results, an optional touch-up application may have been made 4 weeks after the first application.

ELIGIBILITY:
Inclusion Criteria:

* Aged greater than or equal to 18 years
* Female or male
* Volunteers in good general health
* Volunteers with soft tissue deficits on mid-face that can be corrected with volume restoration
* Volunteers who evaluated by investigator as suitable for hyaluronic acid filler applications on her/his lips, nasolabial folds, temporal, perioral, periocular areas
* Individuas who have not filler, botulinum toxin, laser, chemical peeling or surgery in the 6 months before the Semical dermal filler application
* No permanent or non-permanent asthetic applications (chemical peeling, dermabrasion, ablative laser application) non-invasive face-lift, botulinum toxin injections, mesotherapy or fat injections after or simultaneously with filler application
* Volunteers who have not had non-resorbable filler applied before
* Volunteers who have complete records regarding the criteria to be evaluated in the study
* Volunteers who do not have heavy and misleading make-up in their before and after photos
* Volunteers who have not made significant lifestyle changes (diet, physical activity, permanent make-up application)
* No exposure to extreme temperatures such as sunlight, UV solarium, laser, extreme cold, sauna, Turkish baths
* All Fitzpatrick skin types

Exclusion Criteria:

* Patients under 18 years of age
* Presence of impairment of wound healing or blood flow
* Known history of allergy to the study product (hyaluronic acid), local anesthetic used (lidocaine) or gran-positive streptococcal proteins
* Presence or history of keloid formation tendency, hypertrophic scar, shromatosis or discoloration
* Skin disease with pronounced skin pigmentation
* Connective tissue disorders
* Coagulation disorders
* Existing inflammation / infection at the injection site
* Frequently recurring facial / labial herpes
* Permanent or semi-permanent tendon, bone and muscle implants near the area to be application
* History of allergy in the mouth area
* Active autoimmune disease or immunosuppressed individuals with immune system problems
* Diabetes mellitus or uncontrolled systemic disease (endocrine, hepatic, renal, cardiac pulmonary or neurological disorders)
* Volunteers with acute inflammatory conditions or infections, active herpes infection or history of chronic and recurrent infections
* Concomitant medications that affect blood circulation (e.g. aspirin, NSAIDs, Vitamin E, topical and systemic corticosteroids, narcotic antidepressants, immunosuppressive drugs; excluding hormonal and contraceptive treatments started before 1 year) and medications and treatments have the potenrial to affect treatment aoutcomes according to the investigator's opinion
* Known alcohol or drug abuse
* Subjects who are pregnant or breasfeeding
* Subjects who have received COVID-19 vaccination within 30 days before dermal filler application
* Epilepsy or porphyria, congenital or idiopathic methemoglebinemia, or glucose-6-phosphate dehydrogenase deficiency
* Analgesic dependence or need for continuous use
* Syphilis or HIV infection
* Subjects who have undergone medication or surgical treatments that may cause significant changes in body weight after dermal filler application (such as bariatric surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female and male volunteers aged 18 and over who had facial filler application with Semical brand hyaluronic acid dermal fillers at the Akdeniz University Hospital Cosmetology Polyclinic
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
GAIS | From baseline to immediately after injection, 3 months, 6 months, 9 months
  Change of Global Aesthetic Improvement Scale evaluated by patient, investigator and independent rater

SECONDARY OUTCOMES:
WSRS | From baseline to immediately after injection, 3 months, 6 months
  Change of Wrinkle Severity Rating Scale (WSRS) evaluated by patient, investigator and independent rater
Satisfaction of volunteer | From baseline to immediately after injection, 3 montsh, 6 months
  Evaluation of before and after results by visual analogue scale
Ease of use | From baseline to immediately after injection, 3 months, 6 months
  Investigator's assessment for ease of use of the product
Injection pain | During injection and 15 minutes after injection
  Pain perception with visual analogue scale (VAs) during and 15 minutes after injection
Adverse events | throughout the entire study
  Tolerability of the application by evaluation of severity and intensity of the adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University Hospital Dermatology Department Cosmetology Clinic, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Not allowed by local regulations